CLINICAL TRIAL: NCT02000635
Title: Study of Decreasing Kinetics of the Leptospiremia During Antibiotic Treatment of Leptospirosis in Martinique
Acronym: Ciné LEPTO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Center of Martinique (Other)
Collaborators: Clinique Antilles-Guyane (Other)
Responsible Party: Sponsor
Other Study IDs: 13/B/16; 2013-A01128-37 (Registry Identifier: ID RCB)
Record Dates: First submitted 2013-11-20; First posted 2013-12-04 (Estimated); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Leptospirosis
MeSH Terms: conditions — Leptospirosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Leptospirosis: Patient with a diagnosis of leptospirosis confirmed by PCR in the five first day
  Interventions: Other: Quantitative PCR performed at H0 , H24, H48 , H72, 7th day and 14th day

INTERVENTIONS:
Other: Quantitative PCR performed at H0 , H24, H48 , H72, 7th day and 14th day

SUMMARY:
The leptospirosis evolves on an endemic mode in French West Indies and its incidence in 2011 was de 61/100 000 inhabitants, 100 times more than the metropolitan France's incidence (0,47/100 000). If cases can arise all year long, periods of heavy rainfall are associated with the arisen of epidemic peaks Clinical presentation of leptospirosis include a wide range of symptoms: the most frequent form is a flu-like syndrome but more severe forms are described as meningitis, uveitis and classical severe presentation such as lung bleedings and liver-kidneys infringement (syndrome of Weil) which constitute the most severe forms of the disease.

Currently , Polymerase chain reaction (PCR) is the only test who can provide a diagnostic confirmation during the first week of development and before the appearance of the first antibody.

If the microagglutination test (MAT) is considered the gold standard test for diagnosis of leptospirosis. However it requires rending samples to the referent National center for the leptospirosis at Pasteur Institute in Paris while the antibodies do not appears until the second week of illness. A second sample is required 15 days after the first one, to confirm the diagnosis.

In clinical practice , the technique of real-time PCR for the detection and quantification of pathogenic Leptospira during the first week of illness . The technique of diagnosis of leptospirosis by real-time PCR has been implemented and tested in 2007 at the University Hospital of Martinique and providing to the clinicians from 2008. The optimal duration of antibiotic therapy has not been studied and experts now recommend for a 7 to 10 days, regardless of the severity of the disease. The evolution of leptospiremia treated patients has not been studied to date.

ELIGIBILITY:
Inclusion Criteria:

* Adults ( more than 18 years)
* Diagnosis of leptospirosis confirmed by PCR in the five first day
* Appeal to one of the hospital departments participating in the research: in emergency room, in complete hospitalization
* Affiliated patients or beneficiaries of a national insurance scheme
* Acceptance to participate in the study and in the proposed follow-up, and signature of the consent signed by the person or by his(her) representative

Exclusion Criteria:

* Test of negative PCR
* Children under age 18
* No possible follow-up after the first visit
* Pregnant patient
* Refusal of participation in the study
* Unaffiliated patients or beneficiaries of a national insurance scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of leptospirosis confirmed
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-12; Primary Completion 2022-06 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Change of concentration of leptospires in the blood during the first 7 days after the recruitment. | At the recruitment, 24 hours, 48 hours 72 hours and the 7th day after the recruitment
  For each patient, 5-6 quantitative PCR will be performed during the treatment at : The inclusion , 24 hours after the recruitment, 48 hours , 72 hours and the 7th day after the recruitment . In case of positive result of the quantitative PCR at the 7th day of treatment, late charge will be made around the 14th day.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Hochedez, MD, Principal Investigator — CHU de Fort de France
Locations (1):
- Chu de Martinique, Fort-de-France, Martinique